CLINICAL TRIAL: NCT03668418
Title: Xenotransplantation of Primary Cancer Samples in Zebrafish Embryos
Acronym: xenoZ
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Pisa (Other)
Collaborators: Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Principal Investigator, Luca Morelli, Principal Investigator, University of Pisa
Other Study IDs: 70213
Record Dates: First submitted 2018-06-19; First posted 2018-09-12 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Liver Cancer; Pancreatic Cancer; Gastric Cancer; Esophageal Cancer; Colo-rectal Cancer; Gall Bladder Cancer; Biliary Tract Cancer
MeSH Terms: conditions — Liver Neoplasms; Pancreatic Neoplasms; Stomach Neoplasms; Esophageal Neoplasms; Colonic Neoplasms; Gallbladder Neoplasms; Biliary Tract Neoplasms | interventions — Fluorouracil; Leucovorin; Antimetabolites; Oxaliplatin; Platinum Compounds; Irinotecan; Camptothecin; Docetaxel; taxane; Cisplatin; Epirubicin; Anthracyclines; Gemcitabine; Taxes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

GROUPS / COHORTS (4):
- Colorectal cancer: Patients operated for colorectal cancer with or without liver metastasis undergoing a chemotherapy treatment after surgery
  Interventions: Drug: Fluorouracil; Drug: Lederfolin; Drug: Oxaliplatin; Drug: Irinotecan
- Esophagus/gastric cancer: Patients operated for esophagus/gastric cancer undergoing a chemotherapy treatment after surgery
  Interventions: Drug: Fluorouracil; Drug: Lederfolin; Drug: Oxaliplatin; Drug: Irinotecan; Drug: Docetaxel; Drug: Cisplatin; Drug: Epirubicin
- Biliary duct cancer: Patients operated for biliary duct cancer undergoing a chemotherapy treatment after surgery
  Interventions: Drug: Fluorouracil; Drug: Lederfolin; Drug: Oxaliplatin; Drug: Cisplatin; Drug: Gemcitabine
- Pancreatic cancer: Patients operated for pancreatic cancer undergoing a chemotherapy treatment after surgery
  Interventions: Drug: Fluorouracil; Drug: Lederfolin; Drug: Oxaliplatin; Drug: Irinotecan; Drug: Gemcitabine; Drug: Nab paclitaxel

INTERVENTIONS:
Drug: Fluorouracil — The enrolled patients after the surgical operation will undergo to the adjuvant chemotherapy treatment
  Other Names: Fluoropyrimidine
Drug: Lederfolin — The enrolled patients after the surgical operation will undergo to the adjuvant chemotherapy treatment
  Other Names: Antimetabolite
Drug: Oxaliplatin — The enrolled patients after the surgical operation will undergo to the adjuvant chemotherapy treatment
  Other Names: Platinum compounds
Drug: Irinotecan — The enrolled patients after the surgical operation will undergo to the adjuvant chemotherapy treatment
  Other Names: Camptothecin
  Groups: Colorectal cancer; Esophagus/gastric cancer; Pancreatic cancer
Drug: Docetaxel — The enrolled patients after the surgical operation will undergo to the adjuvant chemotherapy treatment
  Other Names: Taxane
  Groups: Esophagus/gastric cancer
Drug: Cisplatin — The enrolled patients after the surgical operation will undergo to the adjuvant chemotherapy treatment
  Other Names: Platinum compounds
  Groups: Biliary duct cancer; Esophagus/gastric cancer
Drug: Epirubicin — The enrolled patients after the surgical operation will undergo to the adjuvant chemotherapy treatment
  Other Names: Anthracycline
  Groups: Esophagus/gastric cancer
Drug: Gemcitabine — The enrolled patients after the surgical operation will undergo to the adjuvant chemotherapy treatment
  Other Names: Antimetabolite
  Groups: Biliary duct cancer; Pancreatic cancer
Drug: Nab paclitaxel — The enrolled patients after the surgical operation will undergo to the adjuvant chemotherapy treatment
  Other Names: Taxane
  Groups: Pancreatic cancer

SUMMARY:
The study consists in a co-clinical trial by using zebrafish embryos. Specifically, an observational prospective clinical trial on patients operated of epato-biliar-pancreatic cancers and gastro-intestinal cancers undergoing a chemotherapy treatment will be run concurrently to an animal trial on zebrafish embryos xenotransplanted with patient cancer cells in order to demonstrate that zebrafish model is able to predict the therapeutic regimen with the best efficacy for each patient.

DETAILED DESCRIPTION:
In the last years, a new concept of personalised medicine called 'Mouse Avatars' or 'co-clinical trials' has emerged. Development of mouse avatars implicates implantation of patient tumour samples in mice for use in drug efficacy studies. This model allows conducting preclinical trials in parallel with ongoing human phase I/II clinical trials. Murine and patient trials are conducted concurrently, and information obtained from the murine system is used for clinical management of the patient's tumour. The advantage of this approach is that each patient has his/her own tumour growing in an in vivo system, thereby allowing the identification of a personalised therapeutic approach. Such approach eliminates the cost and toxicity associated with non-targeted chemotherapy. Unfortunately, nowadays, it is clear that co-clinical trials using mouse avatars are not affordable because mice are expensive and time-consuming. The study challenge is to make Avatars available for every patient and the approach sustainable for the National Healthcare Systems. To implement this concept, the investigators propose to replace mouse Avatars with zebrafish Avatars. Indeed, the investigators propose to run co-clinical trials by using zebrafish embryos. Zebrafish embryos as model for human cancer cell xenografts offer several advantages:

1. Rejection-free model. In zebrafish thymus is not working until 9 days post-fertilization (dpf), allowing rejection-free xenografts during this period. Indeed, the use of expensive immune-permissive strains is not required, in sharp contrast to the mouse model.
2. Very low cost of husbanding.
3. Reduced amount of testing material. Zebrafish experiments require much less material to assess drug efficacy.
4. Short time for the analysis of xenotransplants. The time required for a drug efficacy study is 5 days, as opposite to several weeks or months in the mouse model.
5. Low experimental cost and simple procedures. The zebrafish produces large number of embryos with each fecundation (hundreds). This provides statistical power to the analysis and facilitates the collection of a large number of data.
6. Low ethical impact. Zebrafish is classified as insentient from fecundation to the time at which embryos become capable of independent feeding (120 hours post fertilization, hpf); therefore, during this time it does not require a license according to the Directive 2010/63/EU.
7. Data collected in zebrafish are relevant to humans. Zebrafish genome is closely related to that of humans. For instance, remarkable similarity in molecular signalling processes, cellular structure, anatomy, and physiology has been observed between zebrafish and other high-order vertebrates, including humans. This accounts for the exponential increase in the use of zebrafish in drug discovery during the last two decades.

Collectively, these points outline the remarkable advantages of the zebrafish Avatar over the mouse Avatar, paving the way for a realistic and cost-sustainable implementation of the co-clinical trials.

Specifically, the aim of the study is to perform an observational prospective clinical trial on patients operated of epato-biliar-pancreatic cancers and gastro-intestinal cancers undergoing a chemotherapy treatment in order to demonstrate that zebrafish Avatar is able to predict the therapeutic regimen with the best efficacy for each patient. To this effect, 120 patients meeting the trial inclusion criteria will be enrolled over a 18 months period. In this study, a fragment of tumor will be taken from the surgical specimen by the pathologist, fragmented and transplanted in the yolk of 48 hpf zebrafish embryos. The effect of different anticancer drugs and/or their combinations on the survival, proliferation and migration of the xenotransplanted cancer cells will be evaluated by exposing the xenotransplanted embryos to fish water modified with the drugs. The chemotherapy regimens to be tested in the xenografted embryos are selected in agreement to the common clinical practice, i.e.:

* fluoropyrimidines, platinum compounds, irinotecan, taxans (docetaxel) in stomach & esophageal cancers
* fluoropyrimidines, platinum compounds, irinotecan, gemcitabine, nab paclitaxel in pancreatic/biliary cancers
* fluoropyrimidines, platinum compounds, irinotecan in colorectal cancers.

Embryos will be analysed 4, 24 and 48 hours post injection (hpi). Primary measures will include:

* cell proliferation
* cell migration
* formation of secondary masses
* induction of neo-angiogenesis

The enrolled patients after the surgical operation will undergo to the adjuvant chemotherapy treatment.

The comparative evaluation undertaken after closure of intake will be based on prospectively collected data on (i) clinical outcome and (ii) chemo-sensitivity data collected in zebrafish model.

ELIGIBILITY:
Inclusion Criteria:

- patients operated of epato-biliar-pancreatic cancers and gastro-intestinal cancers (stage III and IV) undergoing a chemotherapy treatment

Exclusion Criteria:

* age below 18 years
* significant co-morbid cardiovascular and respiratory disease
* early stage of disease, (iv) history of prior cancer or prior treatment with any chemotherapy regimen
* pregnant and lactating females
* patients requiring urgent/ emergency interventions
* life expectancy < 12 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Oncological patients from Azienda Ospedaliero-Universitaria Pisana
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Correspondence with chemo-sensitivity data collected in zebrafish model | 18 months after the surgery
  Comparative evaluation between prospectively collected data on clinical outcome and chemo-sensitivity data collected in zebrafish model

SECONDARY OUTCOMES:
Response rate | 3 months after the surgery
  * Complete response (CR) - complete disappearance of clinical evidence of a tumour. Radiographically equivocal lesions must remain stable or regress.
  * Partial response (PR) - 50% or greater decrease in the sum of products of the longest perpendicular diameters of measured lesion compared to baseline.
  * Stable disease (SD) - no significant change in disease status. Lesion may show a <50% decrease in sum of products of longest perpendicular diameters or an increase of <25%.
  * Progressive disease (PD) - a 25% increase in area of a lesion. Appearance of new lesions constitutes progressive disease.
Overall survival | 3 months after the surgery
  The length of time from the start of treatment for the cancer that patients diagnosed with the disease are still alive
Time to tumour progression | 3 months after the surgery
  The length of time from the date of start of treatment for the disease until the disease starts to get worse or spread to other parts of the body
Response rate | 6 months after the surgery
  * Complete response (CR) - complete disappearance of clinical evidence of a tumour. Radiographically equivocal lesions must remain stable or regress.
  * Partial response (PR) - 50% or greater decrease in the sum of products of the longest perpendicular diameters of measured lesion compared to baseline.
  * Stable disease (SD) - no significant change in disease status. Lesion may show a <50% decrease in sum of products of longest perpendicular diameters or an increase of <25%.
  * Progressive disease (PD) - a 25% increase in area of a lesion. Appearance of new lesions constitutes progressive disease.
Overall survival | 6 months after the surgery
  The length of time from the start of treatment for the cancer that patients diagnosed with the disease are still alive
Time to tumour progression | 6 months after the surgery
  The length of time from the date of start of treatment for the disease until the disease starts to get worse or spread to other parts of the body
Response rate | 12 months after the surgery
  * Complete response (CR) - complete disappearance of clinical evidence of a tumour. Radiographically equivocal lesions must remain stable or regress.
  * Partial response (PR) - 50% or greater decrease in the sum of products of the longest perpendicular diameters of measured lesion compared to baseline.
  * Stable disease (SD) - no significant change in disease status. Lesion may show a <50% decrease in sum of products of longest perpendicular diameters or an increase of <25%.
  * Progressive disease (PD) - a 25% increase in area of a lesion. Appearance of new lesions constitutes progressive disease.
Overall survival | 12 months after the surgery
  The length of time from the start of treatment for the cancer that patients diagnosed with the disease are still alive
Time to tumour progression | 12 months after the surgery
  The length of time from the date of start of treatment for the disease until the disease starts to get worse or spread to other parts of the body
Response rate | 18 months after the surgery
  * Complete response (CR) - complete disappearance of clinical evidence of a tumour. Radiographically equivocal lesions must remain stable or regress.
  * Partial response (PR) - 50% or greater decrease in the sum of products of the longest perpendicular diameters of measured lesion compared to baseline.
  * Stable disease (SD) - no significant change in disease status. Lesion may show a <50% decrease in sum of products of longest perpendicular diameters or an increase of <25%.
  * Progressive disease (PD) - a 25% increase in area of a lesion. Appearance of new lesions constitutes progressive disease.
Overall survival | 18 months after the surgery
  The length of time from the start of treatment for the cancer that patients diagnosed with the disease are still alive
Time to tumour progression | 18 months after the surgery
  The length of time from the date of start of treatment for the disease until the disease starts to get worse or spread to other parts of the body

CONTACTS AND LOCATIONS:
Overall Officials: Luca Morelli, Prof, Principal Investigator — University of Pisa
Locations (1):
- Azienda Ospedaliero-Universitaria Pisana, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Usai A, Di Franco G, Piccardi M, Cateni P, Pollina LE, Vivaldi C, Vasile E, Funel N, Palmeri M, Dente L, Falcone A, Giunchi D, Massolo A, Raffa V, Morelli L. Zebrafish Patient-Derived Xenografts Identify Chemo-Response in Pancreatic Ductal Adenocarcinoma Patients. Cancers (Basel). 2021 Aug 17;13(16):4131. doi: 10.3390/cancers13164131. PMID 34439284
- [Derived] Usai A, Di Franco G, Colucci P, Pollina LE, Vasile E, Funel N, Palmeri M, Dente L, Falcone A, Morelli L, Raffa V. A Model of a Zebrafish Avatar for Co-Clinical Trials. Cancers (Basel). 2020 Mar 13;12(3):677. doi: 10.3390/cancers12030677. PMID 32183229